CLINICAL TRIAL: NCT01903187
Title: Multi-center, Randomized, Single-blind, Sham Controlled Clinical Investigation of Renal Denervation for Uncontrolled Hypertension
Brief Title: EnligHTN IV Trial - Multicenter Sham-controlled RCT of Renal Denervation for Hypertension
Acronym: EnligHTN-IV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There were no safety or effectiveness concerns. There were concerns about completing enrollment due to a competitive device's potential approval.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1204
Record Dates: First submitted 2013-07-09; First posted 2013-07-19 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Hypertension
Keywords: hypertension; resistant hypertension; renal denervation
MeSH Terms: conditions — Hypertension | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation (Experimental): Renal artery ablation with the EnligHTN™ Renal Denervation System.
  Interventions: Device: EnligHTN Renal Denervation
- Sham procedure (Active Comparator): Sham procedure
  Interventions: Procedure: Sham

INTERVENTIONS:
Device: EnligHTN Renal Denervation — Renal artery angiogram plus bilateral renal denervation with the EnligHTN renal denervation system
  Arms: Renal Denervation
Procedure: Sham — Renal artery angiogram
  Arms: Sham procedure

SUMMARY:
The purpose of the EnligHTN IV clinical investigation is to demonstrate the safety and effectiveness of the EnligHTN™ Renal Denervation System in the treatment of subjects with drug-resistant uncontrolled hypertension.

DETAILED DESCRIPTION:
The study enrollment was terminated early by the sponsor. This was not related to any safety issue. At the time enrollment was halted, only 2 treatment group randomizations had occurred, and sham group subjects were exited after their 1 month follow up visit.

Subject randomized to the treatment group will be followed up for three years post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age and ≤ 80 years of age at time of informed consent for participation in the clinical investigation
* Subject must be able and willing to provide written informed consent
* Subject must be able and willing to comply with the required follow-up schedule
* Subject has an office Systolic Blood Pressure ≥ 160 mmHg based on an average of 3 Blood Pressure readings at the confirmatory visit (except for subjects with Diabetes Mellitus Type II who must demonstrate an office Systolic Blood Pressure of ≥ 150 mmHg)
* Subject has a daytime mean Systolic 24-hour Ambulatory Blood Pressure value of ≥ 140 mmHg as measured during the two week screening period and confirmed at the confirmatory visit
* Subject is taking ≥ 3 antihypertensive medications concurrently at full tolerated doses (this must include one diuretic) or subject is taking a diuretic and has a documented intolerance to at least two (2) out of the three (3) remaining major classes of anti-hypertensives (ACE / ARB, Calcium Channel Blockers, Beta blockers and is unable to take 3 anti-hypertensive drugs)

  o Intolerance is defined as an absolute contraindication to an anti-hypertensive medication according to the approved labeling or an inability to take an anti-hypertensive medication as prescribed due to an adverse drug effect including an immune mediated response or interaction with other medications.
* Subjects must be on a stable antihypertensive medication regimen for a minimum of 2 weeks prior to completing the initial screening visit and the medication regimen must remain unchanged during the 2 week screening period following signing consent. Subject must be assessed at the confirmatory visit with no expected changes for at least six (6) months

Exclusion Criteria:

* Subject has had a previous renal denervation attempt
* Subject has known cause of secondary hypertension other than sleep apnea
* Subjects with significant renovascular abnormalities such as renal artery stenosis >30%, previous renal stenting or angioplasty, renal artery occlusion, renal vein thrombosis, renal aneurysm or renal atheroembolism
* Subject has had a myocardial infarction, unstable angina pectoris, or cerebrovascular accident < 180 days prior to enrollment
* Subject has hemodynamically significant valvular heart disease as determined by a Study Investigator
* Subject is expected to have any cardiovascular intervention within 180 days of enrollment
* Subject has blood clotting abnormalities such as thrombocytopenia, hemophilia, or significant anemia
* Subject life expectancy is < 12 months, as determined by a Study Investigator
* Subject is participating in another Clinical Investigation (IND or IDE)
* Subject is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods
* Subject has active systemic infection as determined by a Study Investigator
* Subject has main renal arteries with diameter(s) < 4 mm in diameter or < 20 mm in length or multiple renal arteries where the main renal arteries supply <75% of the kidney
* Subject has eGFR < 45 mL/min per 1.73 m2 using the MDRD formula
* Subject has evidence of significant AAA defined as an aneurysm size of ≥5.0 cm in width and/or involving the renal arteries, and/or requiring surgical or percutaneous intervention within 6 months of enrollment.
* Subject has had >1 in-patient hospitalization for a hypertensive crisis within 12 months
* Subject has a condition which would interfere with the accurate interpretation of the study endpoints
* Any condition that would prohibit or interfere with the ability to obtain accurate Blood Pressure measurements using the CIP specific automatic Blood Pressure monitor
* Subject has Systolic Blood Pressure values which are greater than 20mmHg apart after six (6) measurements as assessed at the confirmatory visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B White, MD, Study Chair — UConn Health; William A Gray, MD, Study Chair — Columbia University
Locations (3):
- United States (3):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Jackson Heart Clinic, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Procedure
Arm/Group | Renal Denervation | Sham Procedure
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: 1 Month
Arm/Group | Renal Denervation | Sham Procedure
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: 3 Month
Arm/Group | Renal Denervation | Sham Procedure
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0
Period: 6 Month
Arm/Group | Renal Denervation | Sham Procedure
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0
Period: 12 Month
Arm/Group | Renal Denervation | Sham Procedure
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Denervation | Sham Procedure | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (8.9) | 60.4 (6.7) | 57.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 172.9 (14.1) | 171.5 (5.4) | 172.2 (8.7)
Weight [Mean (Standard Deviation); unit: kilograms] | 81.0 (18.4) | 108.0 (25.0) | 94.5 (23.7)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 27.9 (10.6) | 36.5 (6.2) | 32.2 (8.7)
Years with hypertension [Mean (Standard Deviation); unit: years] | 30.5 (0.7) | 36.0 (0) | 32.3 (3.2)
Coronary Artery Disease [Number; unit: participants]
  Yes | 1 | 0 | 1
  No | 1 | 2 | 3
Renal Artery Stenosis [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 2 | 2 | 4
Hyperlipidemia [Number; unit: participants]
  Yes | 1 | 2 | 3
  No | 1 | 0 | 1
Type II Diabetes [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 2 | 2 | 4
Obstructive Sleep Apnea [Number; unit: participants]
  Yes | 0 | 1 | 1
  No | 2 | 1 | 3
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m2] — Estimated glomular filtration rate use Modified Diet in Renal Disease formula:
  For creatinine in µmol/L:
  eGFR = 32788 X Serum Creatinine^-1.154 X Age^-0.203 X [1.210 if Black] X [0.742 if Female]
  mL/min/1.73 m2 | 91.0 (26.9) | 71.5 (14.8) | 81.3 (21.0)
Serum Creatinine [Mean (Standard Deviation); unit: umol/L] | 69.0 (26.9) | 83.0 (1.4) | 76.0 (17.5)
Cystatin C [Mean (Standard Deviation); unit: mg/L] | 0.76 (0.25) | 0.98 (0.18) | 0.87 (0.22)
Urine Albumin to Creatinine Ratio [Mean (Standard Deviation); unit: mg/g] — Ratio reported as milligrams of albumin per gram of creatinine.
  mg/g | 10.5 (2.1) | 98.0 (106.1) | 54.3 (79.4)
Office Systolic BP [Mean (Standard Deviation); unit: mmHg] | 178.0 (17.0) | 199.5 (34.6) | 188.8 (25.5)
Office Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 111.5 (4.9) | 88.0 (1.4) | 99.8 (13.9)
Office Heart Rate [Mean (Standard Deviation); unit: beats/minute] | 76.5 (12.0) | 58.5 (7.8) | 67.5 (13.3)
24-Hr Ambulatory Systolic BP [Mean (Standard Deviation); unit: mmHg] | 151.7 (22.9) | 155.3 (4.3) | 153.5 (13.6)
24-Hr Ambulatory Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 92.5 (24.7) | 75.4 (1.4) | 83.9 (17.4)
24-Hr Ambulatory Heart Rate [Mean (Standard Deviation); unit: beats/minute] | 68.2 (2.9) | 60.5 (16.0) | 64.3 (10.4)
Daytime Ambulatory Systolic BP [Mean (Standard Deviation); unit: mmHg] | 161.4 (27.0) | 155.0 (2.7) | 158.2 (16.1)
Daytime Ambulatory Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 99.8 (27.6) | 75.6 (1.8) | 87.7 (21.2)
Daytime Ambulatory Heart Rate [Mean (Standard Deviation); unit: beats/minute] | 69.4 (1.6) | 60.6 (18.3) | 65.0 (11.7)
Number of Anti-hypertensive medications [Mean (Standard Deviation); unit: number of anti-hypertensive medications] | 4.0 (1.4) | 5.5 (0.7) | 4.8 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint Will be the Proportion of Subjects Who Experience Any Major Adverse Event (MAE) as Adjudicated by the Clinical Event Committee (CEC).
Description: The study enrollment was terminated early by the sponsor. This was not related to any safety issue. At the time enrollment was halted, only 2 treatment group randomizations had occurred.
Time Frame: 6 months post randomization
Population: All subjects randomized to the EnligHTN procedure
Measure: Number; unit: percentage of participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 2
percentage of participants
  Proportion of Subjects with MAE | 0
  Proportion Subjects without MAE | 100

2. Primary Outcome: The Primary Effectiveness Endpoint is the Reduction of Office Systolic Blood Pressure (OSBP) at Six (6) Months Post Randomization Compared to Baseline Between Groups
Time Frame: 6 months post randomization
Population: The study enrollment was terminated early by the sponsor. This was not related to any safety issue. At the time enrollment was halted, only 2 treatment group randomizations had occurred, and sham group subjects were exited after their 1 month follow up visit. This was not enough to conduct a comparison between groups.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 2 | 0
mmHg | -22.5 (36) |

3. Secondary Outcome: Device or Procedure Related Adverse Events by Severity Post Randomization Through Six (6) Months
Description: The study enrollment was terminated early by the sponsor. This was not related to any safety issue. At the time enrollment was halted, only 2 treatment group randomizations had occurred, and sham group subjects were exited after their 1 month follow up visit. This was not enough to conduct the analysis.
Time Frame: 6 months post randomization
Population: Subjects who received renal denervation
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 2
Participants | 0

4. Secondary Outcome: The Number of Subjects That Experience Each Type of MAE
Description: as for outcome 3
Time Frame: 6 months post randomization
Population: Subjects who received renal denervation
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 2
Participants
  All Cause Mortality | 0
  End Stage Renal Disease (eGFR <15ml/min/m2) | 0
  Significant Embolic Event | 0
  Renal Artery Perforation | 0
  Renal Artery Dissection | 0
  Vascular Access Site Complication | 0
  Hypertensive Crisis | 0
  Renal Artery Stenosis | 0

5. Secondary Outcome: Incidence of Achieving ≥ 10 mmHg, ≥ 15 mmHg, and ≥20 mmHg Reductions in OSBP
Description: as for outcome 3
Time Frame: 6 months post randomization, and all follow-up timepoints
Population: Subjects who received renal denervation
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 2
Participants
  Responders ≥10mmHg SBP reduction from BL(6M) | 1
  Responders ≥10mmHg SBP reduction from BL(12M) | 1
  Responders ≥10mmHg SBP reduction from BL(18M) | 1
  Responders ≥10mmHg SBP reduction from BL(24M): number analyzed (Participants) | 1
  Responders ≥10mmHg SBP reduction from BL(24M) | 1
  Responders ≥10mmHg SBP reduction from BL(30M): number analyzed (Participants) | 1
  Responders ≥10mmHg SBP reduction from BL(30M) | 1
  Responders ≥10mmHg SBP reduction from BL(36M): number analyzed (Participants) | 1
  Responders ≥10mmHg SBP reduction from BL(36M) | 1
  Responders ≥15mmHg SBP reduction from BL (6M) | 1
  Responders ≥15mmHg SBP reduction from BL (12M) | 1
  Responders ≥15mmHg SBP reduction from BL (18M) | 1
  Responders ≥15mmHg SBP reduction from BL (24M): number analyzed (Participants) | 1
  Responders ≥15mmHg SBP reduction from BL (24M) | 1
  Responders ≥15mmHg SBP reduction from BL (30M): number analyzed (Participants) | 1
  Responders ≥15mmHg SBP reduction from BL (30M) | 1
  Responders ≥15mmHg SBP reduction from BL (36M): number analyzed (Participants) | 1
  Responders ≥15mmHg SBP reduction from BL (36M) | 1
  Responders ≥20mmHg SBP reduction from BL (6M) | 1
  Responders ≥20mmHg SBP reduction from BL (12M) | 1
  Responders ≥20mmHg SBP reduction from BL (18M) | 1
  Responders ≥20mmHg SBP reduction from BL (24M): number analyzed (Participants) | 1
  Responders ≥20mmHg SBP reduction from BL (24M) | 1
  Responders ≥20mmHg SBP reduction from BL (30M): number analyzed (Participants) | 1
  Responders ≥20mmHg SBP reduction from BL (30M) | 1
  Responders ≥20mmHg SBP reduction from BL (36M): number analyzed (Participants) | 1
  Responders ≥20mmHg SBP reduction from BL (36M) | 1

6. Secondary Outcome: Reduction in Ambulatory Blood Pressure (ABP) Parameters
Description: as for outcome 3
Time Frame: baseline, 6 months post randomization, and all follow-up timepoints
Population: All subjects
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Sham: Renal artery angiogram without renal denervation
Arm/Group | Renal Denervation | Sham
Number analyzed (Participants) | 2 | 2
mmHg
  Baseline 24Hr Systolic | 151.7 (22.9) | 155.3 (4.3)
  1 Month 24Hr Systolic | 128.8 (1.3) | 155.5 (6.8)
  3 Month 24Hr Systolic: number analyzed (Participants) | 2 | 0
  3 Month 24Hr Systolic | 158.9 (50.8) |
  6 Month 24Hr Systolic: number analyzed (Participants) | 1 | 0
  6 Month 24Hr Systolic | 124.7 (NA) — Cannot calculate standard deviation with one value |
  12 Month 24Hr Systolic: number analyzed (Participants) | 1 | 0
  12 Month 24Hr Systolic | 121.3 (NA) — Cannot calculate standard deviation with one value |
  18 Month 24Hr Systolic: number analyzed (Participants) | 1 | 0
  18 Month 24Hr Systolic | 133.6 (NA) — Cannot calculate standard deviation with one value |
  24 Month 24Hr Systolic: number analyzed (Participants) | 1 | 0
  24 Month 24Hr Systolic | 123.1 (NA) — Cannot calculate standard deviation with one value |
  30 Month 24Hr Systolic: number analyzed (Participants) | 1 | 0
  30 Month 24Hr Systolic | 123.2 (NA) — Cannot calculate standard deviation with one value |
  36 Month 24Hr Systolic: number analyzed (Participants) | 1 | 0
  36 Month 24Hr Systolic | 121.5 (NA) — Cannot calculate standard deviation with one value |
  Baseline 24Hr Diastolic | 92.5 (24.7) | 75.4 (1.4)
  1 Month 24Hr Diastolic | 78.8 (13.5) | 73.9 (4.9)
  3 Month 24Hr Diastolic: number analyzed (Participants) | 2 | 0
  3 Month 24Hr Diastolic | 93.9 (37.8) |
  6 Month 24Hr Diastolic: number analyzed (Participants) | 2 | 0
  6 Month 24Hr Diastolic | 66.2 (NA) — Cannot calculate standard deviation with one value |
  12 Month 24Hr Diastolic: number analyzed (Participants) | 2 | 0
  12 Month 24Hr Diastolic | 67.3 (NA) — Cannot calculate standard deviation with one value |
  18 Month 24Hr Diastolic: number analyzed (Participants) | 2 | 0
  18 Month 24Hr Diastolic | 71.7 (NA) — Cannot calculate standard deviation with one value |
  24 Month 24Hr Diastolic: number analyzed (Participants) | 2 | 0
  24 Month 24Hr Diastolic | 65.2 (NA) — Cannot calculate standard deviation with one value |
  30 Month 24Hr Diastolic: number analyzed (Participants) | 2 | 0
  30 Month 24Hr Diastolic | 61.3 (NA) — Cannot calculate standard deviation with one value |
  36 Month 24Hr Diastolic: number analyzed (Participants) | 2 | 0
  36 Month 24Hr Diastolic | 62.4 (NA) — Cannot calculate standard deviation with one value |

ADVERSE EVENTS:
Time Frame: Ongoing through 3 years post procedure
Description: All events were adjudicated by an independent Clinical Events Committee. Current events included through last annual report (April 2015)
Groups:
- Sham Procedure: Sham procedure
  Sham: Renal artery angiogram
  Subjects exited after 1 month follow up
Arm/Group | Renal Denervation | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=2) | Sham Procedure (N=2)
Subarachnoid Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=2) | Sham Procedure (N=2)
Kidney/Flank Pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhoids/Piles (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other Vascular (Vascular disorders) | 1 (2) | 0 (0) — findings of non-significant plaque or calcium in arteries - unrelated per independent CEC
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment ended early due to a sponsor decision unrelated to safety. The 2 treatment group subjects are being followed up through 3 years. The 2 sham group subjects were exited after their 1 month visit. Due to these reasons, data is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No